CLINICAL TRIAL: NCT01854736
Title: Molecular and Cellular Mechanism in the Course of Immunotherapy With a Phleum Pratense Oral Lyophilisate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GT-24; 2012-005092-14 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-15 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Allergic Rhinitis Due to Grass Pollens
Keywords: Allergy; Phleum pratense; Rhinoconjunctivitis; asthma; positive SPT to Phleum pratense
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Grazax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRAZAX (Active Comparator): Tablet 75.000SQ-T once daily
  Interventions: Drug: Grazax
- Placebo (Placebo Comparator): Tablet with no active grass component
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Grazax — GRAZAX
  Arms: GRAZAX
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This trial is an exploratory randomised, parallel-group, double-blind, placebo- controlled, national, single-centre trial.

The trial will be initiated before 2013 grass pollen season and subjects will be randomised in September 2013 to receive active treatment (Grazax®) or placebo during 2 years. Placebo group will be treated 2 years with placebo and a third year with active therapy (Grazax®) and active group will continue the active treatment in the third year. In the last year, all placebo patients will be changed to active group and active and placebo patients will be informed about, but the trial will not be unblinded until the end of the third year and patients won´t know what treatment they were assigned to during the first 2 years.

DETAILED DESCRIPTION:
There is a first stage of clinical trial (GT-20) in which ALK- Abelló is directly working into the MEICA project to explore human immunological mechanisms of SIT (observed after Grazax® treatment). In this trial, different potential biomarkers of early and sustained effect of specific immunotherapy have been identified. Therefore, for a further research, it was necessary to carry on a new clinical double blind placebo control trial to evaluate a selected panel of biomarkers that can be applied in the selection and monitoring of patients during immunotherapy. They can be of value in the evaluation of future product candidates for specific immunotherapy. For this purpose, it is necessary that the Biomarkers selected, clearly differentiate between active and placebo treated groups. Moreover, specific immunological changes differences between active and placebo patients during pollen seasons are unknown. This first study allowed us identifying a potential set of biomarkers and time points for each of them that might correlate with treatment effect. This second study is needed to evaluate the potential of these biomarkers to discriminate placebo treated patients and it is a necessary step before incorporating them in big prospective efficacy studies.

A third year in an active IMP design after the two years in a double blind placebo setup is included as a way to validate the differences observed intergroup during the first year of therapy. This is needed as pollen seasons significantly differ in strength and duration. Moreover, there is a unique opportunity of analysing immunological changes of the intervention before a careful baseline monitoring of patients undergoing placebo treatment, with the opportunity of understanding immunological clues in the natural evolution of allergy disease.

ELIGIBILITY:
Inclusion Criteria:

* A history of grass pollen allergy
* Positive skin prick test to grass
* Positive specific IgE against Phl p 5
* Written informed consent before entering the trial.
* Female subjects who are fertile must have a negative pregnancy test and be willing to practise appropriate contraceptive methods.
* Subject willing and able to comply with the trial protocol.

Exclusion Criteria:

* Previous treatment by immunotherapy with grass allergen extracts.
* Ongoing treatment with any allergen specific immunotherapy product.
* Previous or ongoing treatment with Omalizumab, mono amine oxidase (MAO) inhibitors or tricyclic antidepressant medication.
* Use of medication at the screening visit which can interfere with SPT results
* A clinical history of symptomatic perennial allergic rhinitis or asthma.
* History of allergy, hypersensitivity or intolerance to the excipients of IMP (except for Phleum pratense).
* Systemic disease affecting the immune system (e.g. autoimmune disease, immune complex disease, or immune deficiency disease).
* Any clinically relevant chronic disease (≥ 3 months duration) (e.g. cystic fibrosis, malignancy, type I diabetes mellitus, malabsorption or malnutrition, renal or hepatic insufficiency).
* Inflammatory conditions in the oral cavity with severe symptoms such as oral lichen planus with ulcerations or severe oral mycosis at randomisation.
* FEV1 ≤ 70% of predicted value.
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process at randomisation.
* Being immediate family of the investigator or trial staff.
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the trial, and/or evidence of an uncooperative attitude.
* Unlikely to be able to complete the trial, for any reason, or likely to move, or travel for extended periods of time during the trial period.
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longest, prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cellular populations (neutrophils, eosinophils, basophils, monocytes, DCs and lymphocytes populations) | 2 years

SECONDARY OUTCOMES:
Global improvement on the Visual Analogue Scale | 2 years
Number of participants with IMP related adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS BLANCO, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (2):
- Spain (2):
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No